CLINICAL TRIAL: NCT06277037
Title: A Long-Term Follow-up Study for Subjects With Chronic Hepatitis B Previously Treated With Imdusiran (AB-729)
Brief Title: Long-Term Follow-up Study for Subjects With CHB Previously Treated With Imdusiran (AB729)
Status: Recruiting | Type: Observational
Sponsor: Arbutus Biopharma Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: AB-729-204
Record Dates: First submitted 2024-02-14; First posted 2024-02-26 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Long Term Follow-up

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Non-interventional — This is a rollover study

SUMMARY:
This is a long term follow-up study for chronic hepatitis B (CHB) subjects who have received imdusiran treatment in a prior clinical trial, stopped NA therapy during that trial, and remain off therapy. Subjects may enroll after completing the end of study visit (baseline visit within 12 weeks ± 1 week from the end of study [EOS] visit) from their imdusiran clinical trial (the "parent study"). No interventions will be performed in this study other than blood sample collections, review of current medications, and reporting of any adverse events related to study procedures or NA therapy if restarted. Study participation will be for approximately 2 years (to complete a total of at least 3 years of follow-up while off NA therapy, inclusive of parent study participation).

ELIGIBILITY:
Key Inclusion Criteria:

* Have participated in a prior imdusiran clinical trial,
* Have discontinued NA therapy in that trial and remain off NA therapy,
* Have completed less than 3 years of follow-up visits after NA discontinuation in the parent study.
* Have the ability to review and provide signed informed consent which includes compliance with all protocol-specified visit schedules and requirements.

Exclusion Criteria:

* Not applicable

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CHB subjects who have received imdusiran treatment in a prior clinical trial, stopped NA therapy during that trial, and remain off therapy at the end of study visit.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-07-11 (Actual); Primary Completion 2029-08-30 (Estimated); Study Completion 2029-10-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the durability of effect of imdusiran on HBV parameters | Up to 96 weeks
  Change from pre-"parent" study baseline and over time in HBsAg, HBV DNA, and hepatitis B surface antibody (HBsAb) at each timepoint.
To evaluate the durability of effect of imdusiran on HBV parameters | Up to 96 weeks
  Proportion of subjects who remain off NA therapy and duration off NA therapy, if applicable
To evaluate the durability of effect of imdusiran on HBV parameters | Up to 96 weeks
  Proportion of subjects who restart NA therapy, if applicable

CONTACTS AND LOCATIONS:
Locations (18):
- United States (3):
  - Research and Education Inc., San Diego, California
  - University of Miami Miller School of Medicine, Miami, Florida
  - Infectious Disease Care, Hillsborough, New Jersey
- Australia (2):
  - The Alfred Hospital, Melbourne, Victoria
  - Fiona Stanley Hospital, Murdoch
- Hong Kong (2):
  - Prince of Wales Hospital, Shatin, New Territories
  - Queen Mary Hospital, Hong Kong
- Arensia Exploratory Medicine Moldova, Chisinau, Moldova
- Asan Medial Center, Seoul, South Korea
- Taiwan (6):
  - Changhua Christian Hospital, Changhua
  - Chia-Yi Christian Hospital, Chiayi City
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - E-Da Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - Chang Gung Medical Foundation Linkou, Taoyuan District
- United Kingdom (3):
  - University Hospital of Wales, Cardiff, Cardiff
  - Royal London Hospital, London
  - King's College Hospital, London

IPD SHARING:
Plan to Share IPD: No